CLINICAL TRIAL: NCT01519817
Title: An Open Label Phase I Study to Evaluate the Safety and Tolerability of GI-6301 Vaccine Consisting of Whole, Heat-Killed Recombinant Saccharomyces Cerevisiae (Yeast) Genetically Modified to Express Brachyury Protein in Adults With Solid Tumors
Brief Title: Cancer Vaccine Targeting Brachyury Protein in Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Senior Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120056; 12-C-0056
Record Dates: First submitted 2012-01-12; First posted 2012-01-27 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Neoplasms; Malignant Solid Tumors; Colon Neoplasms; Adenocarcinoma
Keywords: Vaccine Therapy; Dose-Limiting Toxicity; Maximum Tolerated Dose; Clinical Response; Immune Response; Cancer; Solid Tumor
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Yeast-Brachyury vaccine (Experimental): Yeast-Brachyury vaccine will be administered subcutaneously at 4 sites on 7 visits, then monthly until patients meet off-treatment criteria.
  Interventions: Biological: GI-6301 (Yeast Brachyury Vaccine)

INTERVENTIONS:
Biological: GI-6301 (Yeast Brachyury Vaccine) — GI-6301 is a heat-killed, recombinant yeast-based vaccine engineered to express the transcription factor, Brachyury. The Brachyury gene is used to transfect the parental yeast strain (S. cerevisiae W303 - a haploid strain with known mutations from wildtype yeast) to produce the final recombinant vaccine product.
  Other Names: Yeast-Brachyury vaccine

SUMMARY:
Background:

- Cancer vaccines are being developed to help teach the body's immune system to attack and destroy cancer cells. A new vaccine being tested targets Brachyury protein. This protein is present in some tumor cells, and it can help tumor cells spread to other parts of the body. Researchers want to see whether the new Brachyury protein vaccine can help treat people with advanced carcinomas.

Objectives:

- To test the safety and effectiveness of a cancer vaccine that targets Brachyury protein in tumor cells.

Eligibility:

* Individuals at least 18 years of age who have advanced cancers that have not responded or are no longer responding to standard treatments.
* Because the vaccine is made with yeast, people with yeast allergies will not be eligible.

Design:

* Participants will be screened with a medical history and physical exam. Imaging studies will be used to examine the cancer. Heart and thyroid function tests will be conducted. Blood and urine samples will also be collected.
* Participants will receive vaccine injections every 2 weeks, for a total of seven visits. After seven visits, if the cancer has shrunk or stopped growing, participants will continue to have the vaccine about once a month.
* Treatment will be monitored with frequent blood tests and imaging studies. Other tests will be given as directed by the study doctors. Some participants will have apheresis to collect additional blood cells for study.
* Participants will continue to receive the vaccine as long the tumor does not start growing again and there are no serious side effects....

DETAILED DESCRIPTION:
Background:

* Vaccines based on recombinant heat inactivated yeast have been shown to be immunogenic and well tolerated in animals and humans.
* Using a computer-based differential display analysis tool to conduct global comparison of expressed sequence tag (EST) clusters in the Unigene database, the gene encoding for the transcription factor Brachyury was identified as highly represented in tumor-derived libraries and rarely observed in normal tissue-derived libraries. By using reverse-transcription followed by polymerase chain reaction (RT-PCR), investigators in the LTIB have identified the overexpression of Brachyury in gastrointestinal, bladder, kidney, ovary, uterus, and testicular carcinomas. Similar studies also found over-expression of Brachyury mRNA in cell lines of lung, colon and prostate cancers, but not in the majority of normal tissues tested, with the exception of expression in the testis, thyroid and low levels of expression in B cells pooled from multiple normal donors.
* Brachyury is a member of the T-box family of transcription factors, characterized by a highly conserved DNA-binding domain designated as T-domain. Data indicates that the transcription factor Brachyury confers on the tumor cells a mesenchymal phenotype, as well as migratory and invasive abilities and enhances tumor cell progression.
* A murine model of MC38 cells engineered to over express human Brachyury gene has demonstrated increased metastatic potential of Brachyury over-expressing MC38 cells.
* Brachyury specific T cells can lyse human cancer cells expressing Brachyury in an MHC restricted manner.
* GI-6301 (Yeast-Brachyury vaccine) has been tested in vitro and in the mouse model. These studies showed Brachyury-specific T cell responses and decreased metastasis in mice treated with vaccine.
* An ongoing study of a Hepatitis B vaccine (GS-4774) using the yeast platform (heat killed Saccharomyces cerevisiae) indicated safety of 80 YU dose (4 injection sites at 20 YU injections per site).

Objectives:

-The primary objectives are to:

* Determine the safety and tolerability of escalating doses of GI-6301 (Yeast-Brachyury vaccine) a heat-killed yeast-based vaccine
* Determine in an expanded cohort if a significant change in Brachyury specific T cells will be detectable post vaccine.

Eligibility:

* Adults with histologically proven metastatic or locally advanced solid tumors for which standard curative or palliative measures are no longer effective. Efforts will be made, as much as possible, to enroll patients with tumor types with known increased expression of Brachyury (such as lung, breast, ovarian, prostate, colorectal, pancreatic or chordoma).
* Adequate organ function as defined by liver, kidney, and hematologic laboratory testing.
* Patients with acquired immune defects, systemic autoimmune disease, concurrent use of steroids, pericardial mass > 1 cm, chronic infections, concurrent tricyclic antidepressant therapy, or allergy to yeast or yeast-based products will be excluded.

Design:

* This is an open label, phase I trial with sequential dose escalation cohorts of patients (3-6 patients per dose cohort) for 3 doses of GI-6301 (Yeast-Brachyury vaccine).
* GI-6301 (Yeast-Brachyury vaccine) will be administered subcutaneously at 4 sites biweekly for 7 visits (day 1, 15, 29, 43, 57, 71, 85), then monthly until patients meet off-study criteria

(patients who have been on study for one year or more and have had stable disease or better (PR, CR) have the option to receive vaccine once every 3 months instead of monthly).

* All patients on a given dose level will have completed 28 days on-study without DLT before enrollment can begin on the next dose level or on the expansion phase (see statistical analysis section).
* Expansion Phase: 10 additional patients will be enrolled on the MTD dose level (or the highest dose level explored in the event that a true MTD is not reached), receiving the same treatment regimen, to assess for immunologic responses and clinical responses.
* Amended dose escalation: 10 patients will be enrolled at an additional dose level (80 YU per dose, 4 injection sites at 20 YU per site) to determine the safety of this dose level.
* Up to 33 total patients may be required to complete enrollment of this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants must meet the following criteria for participation:

* Diagnosis: Patients must have histologically confirmed malignancy by the Laboratory of Pathology, National Cancer Institute (NCI), that is metastatic or unresectable locally advanced malignant solid tumor. In the case of Chordoma, unresectable, locally recurrent, or metastatic tumors are acceptable for enrollment, given that this represents incurable disease. Efforts will be made, as much as possible, to enroll patients with tumor types with known increased expression of Brachyury (such as lung, breast, ovarian, prostate, colorectal, pancreatic, or chordoma).
* Patients may have disease that is measurable or non-measurable but evaluable disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at study entry (Karnofsky greater than or equal to 70)
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of Yeast Brachyury vaccine in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Prior Therapy: Completed or had disease progression on at least one prior line of diseaseappropriate therapy for metastatic disease, or not be a candidate for therapy of proven efficacy for their disease.
* Patients must have normal organ and marrow function as defined below:

  * Serum creatinine 1.5 times upper limit of normal OR creatinine clearance on a 24-h urine collection of 60 mL/min.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) 2.5 times the upper limits of normal.
  * Total bilirubin less than or equal to 1.5 times upper limit of normal OR in patients with Gilbert's syndrome, a total bilirubin 3.0.
  * Hematological eligibility parameters (within16 days of starting therapy):
  * Granulocyte count 1,500/mm(3)
  * Platelet count 100,000/m(3)
  * Patients must have baseline pulse oximetry > 90% on room air.
* Recovered completely (Grade 1 or baseline) from any reversible toxicity associated with recent therapy. Typically this is 3 4 weeks for patients who most recently received cytotoxic therapy, except for the nitrosoureas and mitomycin C for which 6 weeks is needed for recovery.
* There should be a minimum of 2 weeks from any prior chemotherapy, immunotherapy and/or radiation.
* Prior immune therapy is allowed.
* Men and women of child-bearing potential must agree to use effective birth control or abstinence during and for a period of 4 months after the last vaccination therapy.
* Patients with prostate cancer must continue to receive gonadotropin-releasing hormone (GnRH) agonist therapy (unless orchiectomy has been done). If a patient has refused GnRH therapy, they may be enrolled on a dose level for which the safety has already been determined.
* Patients with estrogen-receptor positive (ER+) breast cancer being treated with adjuvant hormonal therapy (selective estrogen receptor modulator or aromatase inhibitor) who have rising tumor markers as evidence of disease progression or metastatic disease on scans may continue on hormonal therapy while being treated with vaccine.
* Patients must be negative for yeast allergy skin test
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

Patients with any of the following will not be eligible for participation in this study:

- Patients should have no evidence of immune dysfunction as listed below.

* Human immunodeficiency virus (HIV) positivity due to the potential for decreased immune response to the vaccine.
* Active autoimmune diseases requiring treatment or a history of autoimmune disease that might be stimulated by vaccine treatment. This requirement is due to the potential risks of exacerbating autoimmunity. However, patients with vitiligo, diabetes mellitus, and hashimoto s thyroiditis on appropriate replacement therapy may be

enrolled.

--Concurrent use of systemic steroids, except for physiologic doses of systemic steroid replacement or local (topical, nasal, or inhaled) steroid use. Limited doses of systemic steroids (e.g., in patients with exacerbations of reactive airway disease or to prevent intravenous (IV) contrast allergic reaction or anaphylaxis in patients who have known contrast allergies) are allowed.

* History of allergy or untoward reaction to yeast-based products (any hypersensitivity to yeast-based products will be excluded).
* Pregnant or breast-feeding women, due to the unknown effects of the Yeast Brachyury vaccine on the fetus or infant.
* Serious intercurrent medical illness which would interfere with the ability of the patient to carry out the treatment program, including, but not limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis.
* Untreated brain metastases (or local treatment of brain metastases within the last 6 months) and or spinal cord metastasis.
* Patients with pericardial masses >1 cm will be excluded.
* Concurrent chemotherapy. (However, the following anti-tumor therapies will be allowed: Trastuzumab for human epidermal growth factor receptor 2 (HER2+) breast cancer and hormonal therapy for breast (e.g., selective estrogen receptor modulators, aromatase inhibitors) and prostate cancer (e.g., GnRH antagonists/agonists or antagonists and androgen receptor antagonists).
* Chronic hepatitis infection, including B and C, because potential immune impairment caused by these disorders may diminish the effectiveness of this immunologic therapy.
* Patients requiring continuous tricyclic antidepressant therapy should be excluded due to the interference with the yeast skin test in creating false negative test results.
* Participation in another interventional clinical trial within 28 days before start of study treatment.
* Any significant disease that, in the opinion of the investigator, may impair the patient s tolerance of study treatment.
* Significant dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-01-05 (Actual); Primary Completion 2016-03-03 (Actual); Study Completion 2016-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baranova AV, Lobashev AV, Ivanov DV, Krukovskaya LL, Yankovsky NK, Kozlov AP. In silico screening for tumour-specific expressed sequences in human genome. FEBS Lett. 2001 Nov 9;508(1):143-8. doi: 10.1016/s0014-5793(01)03028-9. PMID 11707285
- [Background] Krukovskaja LL, Baranova A, Tyezelova T, Polev D, Kozlov AP. Experimental study of human expressed sequences newly identified in silico as tumor specific. Tumour Biol. 2005 Jan-Feb;26(1):17-24. doi: 10.1159/000084182. Epub 2005 Feb 28. PMID 15741768
- [Background] Palena C, Polev DE, Tsang KY, Fernando RI, Litzinger M, Krukovskaya LL, Baranova AV, Kozlov AP, Schlom J. The human T-box mesodermal transcription factor Brachyury is a candidate target for T-cell-mediated cancer immunotherapy. Clin Cancer Res. 2007 Apr 15;13(8):2471-8. doi: 10.1158/1078-0432.CCR-06-2353. PMID 17438107
- [Result] Heery CR, Singh BH, Rauckhorst M, Marte JL, Donahue RN, Grenga I, Rodell TC, Dahut W, Arlen PM, Madan RA, Schlom J, Gulley JL. Phase I Trial of a Yeast-Based Therapeutic Cancer Vaccine (GI-6301) Targeting the Transcription Factor Brachyury. Cancer Immunol Res. 2015 Nov;3(11):1248-56. doi: 10.1158/2326-6066.CIR-15-0119. Epub 2015 Jun 30. PMID 26130065
- [Derived] Fenerty KE, Patronas NJ, Heery CR, Gulley JL, Folio LR. Resources Required for Semi-Automatic Volumetric Measurements in Metastatic Chordoma: Is Potentially Improved Tumor Burden Assessment Worth the Time Burden? J Digit Imaging. 2016 Jun;29(3):357-64. doi: 10.1007/s10278-015-9846-9. PMID 26596767
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0056.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 4 YU (Dose Level 1); 16 YU (Dose Level 2); 40 YU (Dose Level 3); 80 YU (Dose Level 4): Yeast-Brachyury vaccine will be administered subcutaneously at 4 sites on 7 visits, then monthly until patients meet off-treatment criteria.
Period: Overall Study
Arm/Group | 4 YU (Dose Level 1) | 16 YU (Dose Level 2) | 40 YU (Dose Level 3) | 80 YU (Dose Level 4)
Started | 4 | 3 | 16 | 11
Completed | 3 | 3 | 16 | 10
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Off study due to infection | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who received at least one dose of 4YU, 16YU, 40YU or 80YU.
  Yeast-Brachyury vaccine will be administered subcutaneously at 4 sites on 7 visits, then monthly until patients meet off-treatment criteria.
  GI-6301 (Yeast Brachyury Vaccine): GI-6301 is a heat-killed, recombinant yeast-based vaccine engineered to express the transcription factor, Brachyury. The Brachyury gene is used to transfect the parental yeast strain (S. cerevisiae W303 - a haploid strain with known mutations from wildtype yeast) to produce the final recombinant vaccine product.
Arm/Group | All Participants
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 58 [32 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 33
  Mexican, Puerto Rican, Cuban Central or So. Americ | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG: 0 is normal activity. Fully active, able to carry on all pre-disease performance without restriction. 1 is symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and bale to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Participants
    0 | 14
    1 | 20
Tumor Type [Count of Participants; unit: Participants]
  Colorectal | 11
  Chordoma | 11
  Breast | 5
  Pancreatic | 3
  Prostate | 2
  Urothelial | 1
  Lung | 1
Disease at Study Entry [Count of Participants; unit: Participants] — Stable disease does not meet criteria for complete response (disappearance of all lesions; no new lesions), partial response (≥30% decrease in the sum of greatest diameters; no new lesions), or progressive disease. Progressive disease is ≥20% increase in the sum of greatest diameters; new lesions. Population: 23 participants with carcinomas (solid tumors) and 11 participants with chordomas.
  Participants
    Carcinomas: number analyzed (Participants) | 23
    Carcinomas: Stable disease | 1
    Carcinomas: Progressive disease | 22
    Chordomas: number analyzed (Participants) | 11
    Chordomas: Stable disease | 2
    Chordomas: Progressive disease | 9
Prior Cytotoxic Regimens [Count of Participants; unit: Participants] — Cytotoxic (i.e. poisonous to cancer cells) Population: The module refers to 23 participants with carcinomas (solid tumors).
  Participants
    0: number analyzed (Participants) | 23
    0 | 1
    1 regimen: number analyzed (Participants) | 23
    1 regimen | 2
    2 regimens: number analyzed (Participants) | 23
    2 regimens | 8
    ≥3 regimens: number analyzed (Participants) | 23
    ≥3 regimens | 12
Tumor Anatomical Location [Count of Participants; unit: Participants] — Sacral (i.e., sacrum), spinal (i.e., backbone), and clival (i.e. base of skull). Population: The module refers to 11 participants with chordomas.
  Participants
    Sacral: number analyzed (Participants) | 11
    Sacral | 6
    Clival: number analyzed (Participants) | 11
    Clival | 3
    Spinal: number analyzed (Participants) | 11
    Spinal | 2
Prior Therapy [Count of Participants; unit: Participants] — Surgery, radiotherapy and systemic therapy use surgical procedures, targeted therapy with radiation, steroids, and/or other immunosuppressive agents in an attempt to suppress one or more growing lesions. Population: The module refers to 11 participants with chordomas.
  Participants
    Surgery: number analyzed (Participants) | 11
    Surgery | 11
    Radiotherapy: number analyzed (Participants) | 11
    Radiotherapy | 11
    Systemic therapy: number analyzed (Participants) | 11
    Systemic therapy | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Brachyury-Specific T-cell Responses
Description: A fluorescense activated cell sorting (FACS)-based assay for cluster of differentiation 4 (CD4) or cluster of differentiation 8 (CD8) T-cells expressing the cytokines interferon (IFN) gamma, interleukin 2 (IL2), and tumor necrosis factor (TNF) alpha, and/or cluster of differentiation 107a (CD107a) (a marker for lytic potential) was used to determine the numbers of participants showing development or enhancement of the level of brachyury-specific T-cells after vaccination.
Time Frame: Baseline (pre-vaccination) and approximately day 84 (after 6 vaccinations)
Population: Sufficient peripheral blood mononuclear cells (PBMCs) were available before and after vaccination from 31 of 34 patients to analyze brachyury-specific CD4 and CD8 T-cell responses.
Measure: Count of Participants; unit: Participants
Arm/Group | 4 YU (Dose Level 1) | 16 YU (Dose Level 2) | 40 YU (Dose Level 3) | 80 YU (Dose Level 4)
Number analyzed (Participants) | 3 | 3 | 16 | 9
Participants
  CD107a + CD4 T-cell response | 1 | 0 | 4 | 1
  IFN gamma + CD4 T-cell response | 1 | 0 | 3 | 2
  IL2 + CD4 T-cell response | 0 | 0 | 3 | 3
  TNF alpha + CD4 T-cell response | 0 | 1 | 6 | 2
  CD107a + CD8 T-cell response | 0 | 0 | 3 | 4
  IFN gamma + CD8 T-cell response | 0 | 0 | 3 | 2
  IL2 + CD8 T-cell response | 0 | 0 | 0 | 1
  TNF alpha + CD8 T-cell response | 0 | 0 | 2 | 3
  Any T-cell response | 1 | 1 | 8 | 7

2. Primary Outcome: Count of Participants With Adverse Events of Escalating Doses of Yeast Brachyury ( GI- 6301) Vaccine
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. A non-serious adverse event is any untoward medical occurrence.
Time Frame: 4 years and 25 days
Measure: Count of Participants; unit: Participants
Arm/Group | 4 YU (Dose Level 1) | 16 YU (Dose Level 2) | 40 YU (Dose Level 3) | 80 YU (Dose Level 4)
Number analyzed (Participants) | 4 | 3 | 16 | 11
Participants | 4 | 3 | 16 | 10

3. Secondary Outcome: Number of Participants With a Clinical Benefit Assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Clinical benefit is defined as partial response (PR) or stable disease (SD) and was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Partial response is ≥30% decrease in the sum of greatest diameters/no new lesions. Progressive disease is ≥20% increase in the sum of greatest diameters/new lesions. Stable disease does not meet criteria for complete response (disappearance of all lesions; no new lesions), partial response, or progressive disease.
Time Frame: 3 and 5 months restaging
Population: One participant was not evaluable and came off study due to infection prior to restaging. Two participants were not evaluable due to withdrawal from the study or lack of measurable disease. Three patients with stable disease at 3 months elected to pursue alternate treatment and did not have 5 month restaging.
Measure: Count of Participants; unit: Participants
Arm/Group | 4 YU (Dose Level 1) | 16 YU (Dose Level 2) | 40 YU (Dose Level 3) | 80 YU (Dose Level 4)
Number analyzed (Participants) | 4 | 3 | 16 | 11
Participants
  Stable disease at 3 months | 3 | 0 | 8 | 6
  Stable disease at 5 months | 2 | 0 | 4 | 3
  Partial response at 3 months | 0 | 0 | 0 | 0
  Partial response at 5 months | 0 | 0 | 1 | 0
  Progressive disease at 3 months | 1 | 3 | 8 | 5
  Progressive disease at 5 months | 1 | 0 | 3 | 0

4. Secondary Outcome: Changes in Immune Cell Subsets in Peripheral Blood Mononuclear Cells (PBMC)
Description: Blood samples will be collected via apheresis and analyzed by multicolor flow cytometry in PBMCs for cluster of differentiation 4 (CD4), cluster of differentiation 8 (CD8), Natural Killer (NK), Natural Killer T (NKT), conventional dendritic cell (cDC), plasmacytoid dendritic cell (pDC), myeloid-derived suppressor cell (MDSC), Tregs, CD4 central memory (CD4 CM), CD4 effector memory (CD4 EM), CD4 terminal effector memory (CD4 EMRA), CD4 naïve, CD8 CM, CD8 EM, CD8 EMRA, and CD8 naïve cells. Significance of changes in immune cells was determined by p value (Wilcoxon test) and the median and interquartile range of data.
Time Frame: Pre (Baseline) and Day 85 after 6 vaccinations
Population: Due to insufficient samples at some time points in some patients, all participants were not analyzed in dose levels 2, 3 and 4; thus a statistical analysis was not performed.
Measure: Median (Inter-Quartile Range); unit: percentage of PBMC
Arm/Group | 4 YU (Dose Level 1) | 16 YU (Dose Level 2) | 40 YU (Dose Level 3) | 80 YU (Dose Level 4)
Number analyzed (Participants) | 4 | 2 | 13 | 9
percentage of PBMC
  Median CD4 Pre | 37.70 [24.11 to 46.36] | 43.57 [40.26 to 46.87] | 29.30 [24.65 to 39.77] | 33.58 [26.84 to 39.92]
  Median CD4 d85 | 38.61 [24.44 to 47.73] | 33.44 [33.37 to 33.52] | 34.29 [25.56 to 37.44] | 27.99 [25.85 to 39.38]
  Median CD8 Pre | 15.87 [8.26 to 16.86] | 14.77 [3.49 to 26.04] | 15.96 [10.76 to 19.48] | 13.76 [10.31 to 19.77]
  Median CD8 d85 | 15.67 [9.102 to 16.57] | 13.63 [4.123 to 23.14] | 15.42 [10.96 to 22.44] | 16.02 [10.57 to 25.5]
  Median B cells Pre | 7.05 [6.19 to 10.07] | 11.02 [9.92 to 12.11] | 8.97 [3.54 to 12.13] | 7.82 [3.13 to 12.07]
  Median B cells d85 | 6.93 [6.16 to 10.58] | 9.78 [7.95 to 11.62] | 9.10 [5.07 to 12.17] | 8.77 [3.78 to 10.72]
  Median Natural Killer (NK) Pre | 5.21 [4.14 to 6.94] | 6.57 [3.27 to 9.87] | 5.72 [3.13 to 8.51] | 5.89 [4.59 to 9.14]
  Median Natural Killer (NK) d85 | 5.72 [4.03 to 7.39] | 8.41 [5.50 to 11.31] | 4.22 [3.97 to 10.07] | 9.14 [5.95 to 11.4]
  Median Natural Killer T cell (NKT) Pre | 1.00 [0.65 to 4.21] | 1.70 [0.46 to 2.94] | 1.27 [0.62 to 2.81] | 2.24 [0.59 to 4.39]
  Median Natural Killer T cell (NKT) d85 | 1.25 [0.67 to 4.75] | 2.46 [0.51 to 4.40] | 1.19 [0.58 to 3.15] | 2.53 [0.77 to 5.86]
  Median cDC Pre | 0.25 [0.14 to 0.28] | 0.14 [0.11 to 0.17] | 0.23 [0.20 to 0.37] | 0.17 [0.16 to 0.35]
  Median cDC d85 | 0.18 [0.14 to 0.23] | 0.17 [0.16 to 0.19] | 0.21 [0.18 to 0.34] | 0.19 [0.09 to 0.23]
  Median pDC Pre | 0.25 [0.20 to 0.37] | 0.17 [0.09 to 0.24] | 0.23 [0.17 to 0.36] | 0.23 [0.11 to 0.31]
  Median pDC d85 | 0.32 [0.27 to 0.38] | 0.26 [0.08 to 0.44] | 0.27 [0.18 to 0.35] | 0.23 [0.14 to 0.40]
  Median MDSC Pre | 10.98 [2.96 to 19.19] | 8.53 [4.30 to 12.76] | 8.47 [5.98 to 14.54] | 13.73 [5.41 to 17.61]
  Median MDSC d85 | 11.41 [4.82 to 18.78] | 10.78 [5.98 to 15.58] | 7.55 [4.95 to 12.16] | 12.77 [6.64 to 14.23]
  Median Treg Pre | 0.77 [0.66 to 0.90] | 0.90 [0.68 to 1.13] | 1.25 [0.73 to 1.74] | 1.07 [0.55 to 1.60]
  Median Treg d85 | 0.81 [0.78 to 1.03] | 0.80 [0.42 to 1.17] | 1.12 [0.83 to 1.71] | 1.00 [0.45 to 1.41]
  Median CD4 EM Pre | 10.58 [8.47 to 12.73] | 12.09 [9.67 to 14.51] | 13.14 [10.67 to 14.82] | 11.31 [8.49 to 15.97]
  Median CD4 EM d85 | 8.92 [7.49 to 13.48] | 10.72 [9.20 to 12.25] | 12.50 [11.33 to 13.63] | 9.76 [7.21 to 15.68]
  Median CD4 CM Pre | 17.29 [8.59 to 21.10] | 23.20 [12.62 to 33.79] | 12.36 [9.16 to 17.44] | 12.07 [7.52 to 16.56]
  Median CD4 CM d85 | 18.80 [9.75 to 24.37] | 16.51 [10.97 to 22.06] | 12.78 [10.53 to 17.98] | 11.36 [6.00 to 14.40]
  Median CD4 EMRA Pre | 0.32 [0.28 to 1.96] | 0.68 [0.21 to 1.15] | 0.34 [0.26 to 0.90] | 0.28 [0.21 to 1.04]
  Median CD4 EMRA d85 | 0.34 [0.26 to 0.70] | 0.83 [0.24 to 1.43] | 0.28 [0.23 to 0.56] | 0.38 [0.21 to 1.75]
  Median CD4 naive Pre | 10.28 [4.23 to 12.36] | 7.57 [3.23 to 11.91] | 3.78 [2.47 to 6.90] | 4.49 [2.56 to 10.22]
  Median CD4 naive d85 | 8.48 [4.14 to 12.76] | 5.41 [2.08 to 8.73] | 3.99 [3.49 to 7.51] | 6.08 [3.15 to 9.55]
  Median CD8 EM Pre | 3.20 [2.33 to 6.85] | 2.70 [1.54 to 3.86] | 7.19 [4.45 to 8.92] | 5.23 [4.21 to 7.64]
  Median CD8 EM d85 | 3.44 [2.85 to 6.87] | 3.33 [2.61 to 4.06] | 6.60 [4.12 to 10.78] | 6.11 [3.91 to 7.30]
  Median CD8 CM Pre | 1.03 [0.61 to 2.70] | 1.05 [0.80 to 1.30] | 1.16 [0.56 to 1.48] | 1.00 [0.53 to 1.38]
  Median CD8 CM d85 | 1.31 [0.81 to 2.43] | 0.86 [0.53 to 1.19] | 0.95 [0.80 to 1.44] | 0.88 [0.32 to 1.26]
  Median CD8 EMRA Pre | 3.01 [1.22 to 8.46] | 2.51 [0.63 to 4.39] | 2.60 [1.36 to 9.95] | 5.81 [2.26 to 8.75]
  Median CD8 EMRA d85 | 2.84 [1.40 to 7.35] | 3.24 [0.69 to 5.80] | 3.31 [1.14 to 10.71] | 5.06 [3.11 to 10.83]
  Median CD8 naive Pre | 3.47 [2.50 to 5.60] | 8.51 [0.53 to 16.49] | 2.43 [0.92 to 5.25] | 3.71 [2.86 to 5.92]
  Median CD8 naive d85 | 3.28 [2.58 to 6.21] | 6.20 [0.30 to 12.09] | 3.12 [1.00 to 5.82] | 3.44 [2.06 to 5.45]
Statistical Analysis 1: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.5221, Wilcoxon test — The reported p-value is representative of the changes in levels of all CD4 cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 2: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.25, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 cells at dose level 1
Statistical Analysis 3: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.50, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 cells at dose level 3
Statistical Analysis 4: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.16, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 cells at dose level 4
Statistical Analysis 5: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.8665, Wilcoxon test — The reported p-value is representative of the changes in levels of all CD8 cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 6: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.88, Wilcoxon test — [p-value comment as in outcome 4, analysis 5]
Statistical Analysis 7: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.84, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 cells at dose level 3
Statistical Analysis 8: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.57, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 cells at dose level 4
Statistical Analysis 9: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.3052, Wilcoxon test — The reported p-value is representative of the changes in levels of all B cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 10: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.9999, Wilcoxon test — The reported p-value is representative of the changes in levels of B cells at dose level 1; The reported p-value is representative of the changes in levels of B cells at dose level 1
Statistical Analysis 11: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.13, Wilcoxon test — The reported p-value is representative of the changes in levels of B cells at dose level 3
Statistical Analysis 12: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.65, Wilcoxon test — The reported p-value is representative of the changes in levels of B cells at dose level 4
Statistical Analysis 13: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.0698, Wilcoxon test — The reported p-value is representative of the changes in levels of all NK cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 14: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.63, Wilcoxon test — The reported p-value is representative of the changes in levels of NK cells at dose level 1
Statistical Analysis 15: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.74, Wilcoxon test — The reported p-value is representative of the changes in levels of NK cells at dose level 3
Statistical Analysis 16: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.13, Wilcoxon test — The reported p-value is representative of the changes in levels of NK cells at dose level 4
Statistical Analysis 17: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.0127, Wilcoxon test — The reported p-value is representative of the changes in levels of all NKT cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 18: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.63, Wilcoxon test — The reported p-value is representative of the changes in levels of NKT cells at dose level 1
Statistical Analysis 19: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.41, Wilcoxon test — The reported p-value is representative of the changes in levels of NKT cells at dose level 3
Statistical Analysis 20: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.07, Wilcoxon test — The reported p-value is representative of the changes in levels of NKT cells at dose level 4
Statistical Analysis 21: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.0654, Wilcoxon test — The reported p-value is representative of the changes in levels of all cDC cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 22: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.38, Wilcoxon test — The reported p-value is representative of the changes in levels of cDC cells at dose level 1
Statistical Analysis 23: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.21, Wilcoxon test — The reported p-value is representative of the changes in levels of cDC cells at dose level 3
Statistical Analysis 24: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.16, Wilcoxon test — The reported p-value is representative of the changes in levels of cDC cells at dose level 4
Statistical Analysis 25: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.0457, Wilcoxon test — The reported p-value is representative of the changes in levels of all pDC cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 26: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.63, Wilcoxon test — The reported p-value is representative of the changes in levels of pDC cells at dose level 1
Statistical Analysis 27: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.55, Wilcoxon test — The reported p-value is representative of the changes in levels of pDC cells at dose level 3
Statistical Analysis 28: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.13, Wilcoxon test — The reported p-value is representative of the changes in levels of pDC cells at dose level 4
Statistical Analysis 29: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.7114, Wilcoxon test — The reported p-value is representative of the changes in levels of all MDSC cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 30: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.9999, Wilcoxon test — The reported p-value is representative of the changes in levels of MDSC cells at dose level 1
Statistical Analysis 31: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.38, Wilcoxon test — The reported p-value is representative of the changes in levels of MDSC cells at dose level 3
Statistical Analysis 32: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.91, Wilcoxon test — The reported p-value is representative of the changes in levels of MDSC cells at dose level 4
Statistical Analysis 33: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.2666, Wilcoxon test — The reported p-value is representative of the changes in levels of all Treg cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 34: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.88, Wilcoxon test — The reported p-value is representative of the changes in levels of Treg cells at dose level 1
Statistical Analysis 35: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.45, Wilcoxon test — The reported p-value is representative of the changes in levels of Treg cells at dose level 1
Statistical Analysis 36: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.36, Wilcoxon test — The reported p-value is representative of the changes in levels of Treg cells at dose level 4
Statistical Analysis 37: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.0076, Wilcoxon test — The reported p-value is representative of the changes in levels of all CD4 EM cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 38: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.38, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 EM cells at dose level 1
Statistical Analysis 39: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.22, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 EM cells at dose level 3
Statistical Analysis 40: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.10, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 EM cells at dose level 4
Statistical Analysis 41: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.7144, Wilcoxon test — The reported p-value is representative of the changes in levels of all CD4 CM cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 42: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.13, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 CM cells at dose level 1
Statistical Analysis 43: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.06, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 CM cells at dose level 3
Statistical Analysis 44: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.13, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 CM cells at dose level 4
Statistical Analysis 45: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.3741, Wilcoxon test — The reported p-value is representative of the changes in levels of all CD4 EMRA cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 46: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — The reported p-value is representative of the changes in levels of CD4 EMRA cells at dose level 1; p = 0.63, Wilcoxon test
Statistical Analysis 47: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.13, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 EMRA cells at dose level 3
Statistical Analysis 48: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.9999, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 EMRA cells at dose level 4
Statistical Analysis 49: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.3386, Wilcoxon test — The reported p-value is representative of the changes in levels of all CD4 naive cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 50: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.88, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 naive cells at dose level 1
Statistical Analysis 51: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.0215, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 naive cells at dose level 3
Statistical Analysis 52: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.65, Wilcoxon test — The reported p-value is representative of the changes in levels of CD4 naive cells at dose level 4
Statistical Analysis 53: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.5076, Wilcoxon test — The reported p-value is representative of the changes in levels of all CD8 EM cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 54: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.63, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 EM cells at dose level 1
Statistical Analysis 55: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.68, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 EM cells at dose level 3
Statistical Analysis 56: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.73, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 EM cells at dose level 4
Statistical Analysis 57: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.6577, Wilcoxon test — The reported p-value is representative of the changes in levels of all CD8 CM cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 58: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.88, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 CM cells at dose level 1
Statistical Analysis 59: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.74, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 CM cells at dose level 3
Statistical Analysis 60: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.20, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 CM cells at dose level 4
Statistical Analysis 61: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.6295, Wilcoxon test — The reported p-value is representative of the changes in levels of all CD8 EMRA cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 62: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.63, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 EMRA cells at dose level 1
Statistical Analysis 63: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.999, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 EMRA cells at dose level 3
Statistical Analysis 64: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.36, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 EMRA cells at dose level 4
Statistical Analysis 65: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.8314, Wilcoxon test — The reported p-value is representative of the changes in levels of all CD8 naive cells at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 66: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — The reported p-value is representative of the changes in levels of CD8 naive cells at dose level 1; p = 0.63, Wilcoxon test
Statistical Analysis 67: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.64, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 naive cells at dose level 3
Statistical Analysis 68: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.30, Wilcoxon test — The reported p-value is representative of the changes in levels of CD8 naive cells at dose level 4

5. Secondary Outcome: Changes in Serum Levels of Cytokines
Description: Blood samples were collected and changes in serum levels of cytokines interferon gamma (IFNg), Interleukin 10 (IL-10), Interleukin 12 (IL-12)p70, Interleukin 1b (IL-1b), Interleukin 2 (IL-2), Interleukin 6 (IL-6), Interleukin 8 (IL-8), and tumor necrosis factor (TNF) were assessed by the multiplexed mesoscale assay. Significance of changes in serum levels of cytokines was determined by p value (Wilcoxon test) and the median and interquartile range of data.
Time Frame: Pre (Baseline) and Day 85 after 6 vaccinations
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | 4 YU (Dose Level 1) | 16 YU (Dose Level 2) | 40 YU (Dose Level 3) | 80 YU (Dose Level 4)
Number analyzed (Participants) | 4 | 2 | 12 | 9
pg/ml
  Median IFNg Pre | 3.63 [2.47 to 6.12] | 3.56 [2.99 to 4.13] | 2.805 [1.97 to 3.6] | 4.47 [4.05 to 7.48]
  Median IFNg d85 | 2.64 [2.17 to 3.17] | 2.83 [2.62 to 3.04] | 2.84 [1.76 to 4.71] | 4.9 [2.91 to 6.81]
  Median IL-10 Pre | 0.24 [0.17 to 0.54] | 0.215 [0.2 to 0.23] | 0.21 [0.17 to 0.28] | 0.4 [0.31 to 0.47]
  Median IL-10 d85 | 0.26 [0.23 to 0.39] | 0.285 [0.28 to 0.29] | 0.24 [0.18 to 0.31] | 0.4 [0.26 to 0.52]
  Median IL-12p70 Pre | 0.2 [0.2 to 0.22] | 0.22 [0.2 to 0.24] | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.37]
  Median IL-12p70 d85 | 0.2 [0.2 to 0.28] | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.2] | 0.2 [0.2 to 0.26]
  Median IL-1b Pre | 0.24 [0.24 to 1.15] | 0.24 [0.24 to 0.24] | 0.24 [0.24 to 0.24] | 0.24 [0.24 to 2.52]
  Median IL-1b d85 | 0.24 [0.24 to 0.25] | 0.24 [0.24 to 0.24] | 0.24 [0.24 to 0.24] | 0.24 [0.24 to 0.89]
  Median IL-2 Pre | 0.64 [0.64 to 2.40] | 0.64 [0.64 to 0.64] | 0.64 [0.64 to 0.64] | 0.64 [0.64 to 0.80]
  Median IL-2 d85 | 0.64 [0.64 to 0.93] | 0.64 [0.64 to 0.64] | 0.64 [0.64 to 0.64] | 0.64 [0.64 to 0.70]
  Median IL-6 Pre | 0.88 [0.71 to 2.85] | 0.78 [0.66 to 0.9] | 1.02 [0.52 to 1.3] | 2.37 [0.69 to 15.3]
  Median IL-6 d85 | 0.97 [0.74 to 1.23] | 0.855 [0.76 to 0.95] | 1.04 [0.54 to 1.97] | 2.84 [0.90 to 4.84]
  Median IL-8 Pre | 56.45 [16.84 to 487.6] | 43.87 [16.05 to 71.69] | 37.49 [18 to 91.01] | 63.52 [33.7 to 560.2]
  Median IL-8 d85 | 33.29 [30.52 to 124.5] | 61.85 [44.98 to 78.71] | 43.27 [17.99 to 140.1] | 73.21 [38.62 to 200.9]
  Median TNF Pre | 1.54 [1.19 to 8.19] | 1.315 [1.24 to 1.39] | 1.62 [1.25 to 2.26] | 3.59 [2.19 to 9.24]
  Median TNF d85 | 1.63 [1.45 to 1.81] | 1.465 [1.23 to 1.7] | 1.67 [1.38 to 2.07] | 2.74 [2.26 to 3.77]
Statistical Analysis 1: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.375, Wilcoxon test — The reported p-value is representative of the changes in levels of IFNg cytokines at dose level 1
Statistical Analysis 2: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.4808, Wilcoxon test — The reported p-value is representative of the changes in levels of all IFNg cytokines at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 3: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.7334, Wilcoxon test — The reported p-value is representative of the changes in levels of IFNg cytokines at dose level 3
Statistical Analysis 4: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.7109, Wilcoxon — The reported p-value is representative of the changes in levels of IFNg cytokines at dose level 4
Statistical Analysis 5: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.4347, Wilcoxon test — The reported p-value is representative of the changes in levels of all IL10 cytokines at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 6: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.9999, Wilcoxon — The reported p-value is representative of the changes in levels of IL10 cytokines at dose level 1
Statistical Analysis 7: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.748, Wilcoxon test — The reported p-value is representative of the changes in levels of IL10 cytokines at dose level 3
Statistical Analysis 8: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.8203, Wilcoxon test; The reported p-value is representative of the changes in levels of IL10 cytokines at dose level 4
Statistical Analysis 9: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.5625, Wilcoxon test — The reported p-value is representative of the changes in levels of all IL12p70 cytokines at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 10: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.9999, Wilcoxon test — The reported p-value is representative of the changes in levels of IL12p70 cytokines at dose level 1
Statistical Analysis 11: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.9999, Wilcoxon test — The reported p-value is representative of the changes in levels of IL12p70 cytokines at dose level 3
Statistical Analysis 12: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.5, Wilcoxon test — The reported p-value is representative of the changes in levels of IL12p70 cytokines at dose level 14
Statistical Analysis 13: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.6846, Wilcoxon test — The reported p-value is representative of the changes in levels of all IL1b cytokines at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 14: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.9999, Wilcoxon test — The reported p-value is representative of the changes in levels of IL1b cytokines at dose level 1
Statistical Analysis 15: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.5, Wilcoxon test — The reported p-value is representative of the changes in levels of IL1b cytokines at dose level 3
Statistical Analysis 16: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.9999, Wilcoxon test — The reported p-value is representative of the changes in levels of IL1b cytokines at dose level 4
Statistical Analysis 17: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.4375, Wilcoxon test — The reported p-value is representative of the changes in levels of all IL-2 cytokines at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 18: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.9999, Wilcoxon test — The reported p-value is representative of the changes in levels of IL-2 cytokines at dose level 1
Statistical Analysis 19: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.9999, Wilcoxon test — The reported p-value is representative of the changes in levels of IL-2 cytokines at dose level 3
Statistical Analysis 20: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.75, Wilcoxon test — The reported p-value is representative of the changes in levels of IL-2 cytokines at dose level 4
Statistical Analysis 21: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.4525, Wilcoxon test — The reported p-value is representative of the changes in levels of all IL-6 cytokines at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses; The reported p-value is representative of the changes in levels of IL-6 cytokines at dose level 1
Statistical Analysis 22: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.875, Wilcoxon test — The reported p-value is representative of the changes in levels of IL-6 cytokines at dose level 1
Statistical Analysis 23: Comparison: 40 YU (Dose Level 3); Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; Test type: Non-Inferiority — The reported p-value is representative of the changes in levels of IL-6 cytokines at dose level 3; p = 0.4316, Wilcoxon test
Statistical Analysis 24: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.9999, Wilcoxon test — The reported p-value is representative of the changes in levels of IL-6 cytokines at dose level 4
Statistical Analysis 25: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.9906, Wilcoxon test — The reported p-value is representative of the changes in levels of all IL-8 cytokines at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 26: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.625, Wilcoxon test; The reported p-value is representative of the changes in levels of IL-8 cytokines at dose level 1
Statistical Analysis 27: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.791, Wilcoxon test — The reported p-value is representative of the changes in levels of IL-8 cytokines at dose level 3
Statistical Analysis 28: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.8203, Wilcoxon test — The reported p-value is representative of the changes in levels of IL-8 cytokines at dose level 4
Statistical Analysis 29: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p > 0.9999, Wilcoxon test — The reported p-value is representative of the changes in levels of all TNF cytokines at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 30: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.875, Wilcoxon test — The reported p-value is representative of the changes in levels of TNF cytokines at dose level 1
Statistical Analysis 31: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.9658, Wilcoxon test — The reported p-value is representative of the changes in levels of TNF cytokines at dose level 3
Statistical Analysis 32: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.6523, Wilcoxon test — The reported p-value is representative of the changes in levels of TNF cytokines at dose level 4

6. Secondary Outcome: Changes in Soluble Cluster of Differentiation 27 (sCD27)
Description: Blood samples were collected and changes in serum levels of soluble sCD27 were assessed by enzyme-linked immunosorbent assay (ELISA). Significance of changes in soluble sCD27 was determined by p value (Wilcoxon test) and the median and interquartile range of data.
Time Frame: Pre (Baseline) and Day 85 after 6 vaccinations
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: U/ml
Arm/Group | 4 YU (Dose Level 1) | 16 YU (Dose Level 2) | 40 YU (Dose Level 3) | 80 YU (Dose Level 4)
Number analyzed (Participants) | 4 | 2 | 12 | 9
U/ml
  Median sCD27 Pre | 99.07 [91.13 to 131] | 98.63 [87.12 to 110.1] | 97.47 [85.15 to 110.9] | 128.4 [123.9 to 145.6]
  Median sCD27 d85 | 97.17 [92.07 to 1112] | 92.07 [83.3 to 100.8] | 101.7 [98.85 to 105.1] | 133.1 [129.7 to 155.8]
Statistical Analysis 1: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.2901, Wilcoxon test — The reported p-value is representative of the changes in levels of all sCD27 cytokines at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 2: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.375, Wilcoxon test — The reported p-value is representative of the changes in levels of sCD27 cytokines at dose level 1
Statistical Analysis 3: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.2036, Wilcoxon test — The reported p-value is representative of the changes in levels of sCD27 cytokines at dose level 3
Statistical Analysis 4: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.0742, Wilcoxon test — The reported p-value is representative of the changes in levels of sCD27 cytokines at dose level 4

7. Secondary Outcome: Median Ratio of Soluble Cluster of Differentiation 27:40L (sCD27:sCD40L)
Description: Blood samples were collected and changes in serum levels of the ratio of soluble sCD27:sCD40L was assessed by enzyme-linked immunosorbent assay (ELISA). Significance of changes in soluble sCD27:sCD40L was determined by p value (Wilcoxon test) and the median and interquartile range of data.
Time Frame: Pre (Baseline) and Day 85 after 6 vaccinations
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | 4 YU (Dose Level 1) | 16 YU (Dose Level 2) | 40 YU (Dose Level 3) | 80 YU (Dose Level 4)
Number analyzed (Participants) | 4 | 2 | 12 | 9
Ratio
  Median sCD27:sCD40L Pre | 5.982 [5.71 to 11.67] | 9.57 [7.88 to 11.26] | 9.571 [7.67 to 19.89] | 8.57 [6.93 to 10.62]
  Median sCD27:sCD40L d85 | 6.428 [4.79 to 9.43] | 8.294 [7.29 to 9.29] | 10.47 [6.63 to 19.38] | 8.257 [6.96 to 8.91]
Statistical Analysis 1: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.1004, Wilcoxon test — The reported p-value is representative of the changes in levels of all ratio sCD27:sCD40AL cytokines at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 2: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.625, Wilcoxon test — The reported p-value is representative of the changes in levels of ratio sCD27:sCD40L cytokines at dose level 1
Statistical Analysis 3: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.6772, Wilcoxon test — The reported p-value is representative of the changes in levels of ratio sCD27:sCD40L cytokines at dose level 3
Statistical Analysis 4: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.3008, Wilcoxon test — The reported p-value is representative of the changes in levels of ratio sCD27:sCD40L cytokines at dose level 4

8. Secondary Outcome: Changes in Soluble Cluster of Differentiation 40L (sCD40L)
Description: Blood samples were collected and changes in serum levels of soluble sCD27 were assessed by enzyme-linked immunosorbent assay (ELISA). Significance of changes in soluble sCD40L was determined by p value (Wilcoxon test) and the median and interquartile range of data.
Time Frame: Pre (Baseline) and Day 85 after 6 vaccinations
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | 4 YU (Dose Level 1) | 16 YU (Dose Level 2) | 40 YU (Dose Level 3) | 80 YU (Dose Level 4)
Number analyzed (Participants) | 4 | 2 | 12 | 9
ng/ml
  Median sCD40L Pre | 15.3 [11.39 to 17.99] | 10.24 [9.78 to 11.06] | 9.648 [5.27 to 13.99] | 14.72 [13.67 to 18.74]
  Median sCD40L d85 | 15.23 [11.96 to 19.42] | 11.14 [10.84 to 11.43] | 9.854 [5.86 to 14.52] | 18.57 [16.09 to 19.51]
Statistical Analysis 1: Comparison: 4 YU (Dose Level 1) vs 40 YU (Dose Level 3) vs 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.0621, Wilcoxon test — The reported p-value is representative of the changes in levels of all sCD40L cytokines at dose levels 1, 3, and 4. We could not do dose level 2 as we only had data on 2 patients and need an n>2 to do paired analyses
Statistical Analysis 2: Comparison: 4 YU (Dose Level 1); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.875, Wilcoxon test — The reported p-value is representative of the changes in levels of sCD40L cytokines at dose level 1
Statistical Analysis 3: Comparison: 40 YU (Dose Level 3); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.2402, Wilcoxon test — The reported p-value is representative of the changes in levels of sCD40L cytokines at dose level 3
Statistical Analysis 4: Comparison: 80 YU (Dose Level 4); Test type: Non-Inferiority — Significance was met if the unadjusted p-value was <0.05 and >1/2 of patients had a serum level change of >25%; p = 0.3008, Wilcoxon test — The reported p-value is representative of the changes in levels of sCD40L cytokines at dose level 4

ADVERSE EVENTS:
Time Frame: 4 years and 25 days
Arm/Group | 4 YU (Dose Level 1) | 16 YU (Dose Level 2) | 40 YU (Dose Level 3) | 80 YU (Dose Level 4)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/16 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 5/16 | 6/11
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 16/16 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 YU (Dose Level 1) (N=4) | 16 YU (Dose Level 2) (N=3) | 40 YU (Dose Level 3) (N=16) | 80 YU (Dose Level 4) (N=11)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, lung obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 YU (Dose Level 1) (N=4) | 16 YU (Dose Level 2) (N=3) | 40 YU (Dose Level 3) (N=16) | 80 YU (Dose Level 4) (N=11)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (4) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 4 (4) | 3 (3)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (6) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 4 (7) | 1 (2) | 0 (0) | 9 (33)
Lymphocyte count decreased (Investigations) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (3) | 0 (0) | 0 (0) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Platelet count decreased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 11 (16) | 3 (7)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 3 (4) | 1 (3)
Skin and subcutaneous tissue disorders - Other,R hand skin mass,excision 11/27/12 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 1 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin I increased (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (3)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 3 (6)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (3) | 4 (4)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (6) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 4 (7) | 0 (0) | 10 (23) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other, hemoglobinuria (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nervous system disorders - Other, lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal disorders - Other, poor appetite (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, nephrostomy tube site (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder-Other, R knee swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — gr. 1, unrelated
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Body aches (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Erythema/redness R LE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, sebac cyst-back (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, R knee redness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, bruised R big toe (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, itching nose intermittent (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, top R foot open wound (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-01-06): https://cdn.clinicaltrials.gov/large-docs/17/NCT01519817/Prot_SAP_ICF_000.pdf